CLINICAL TRIAL: NCT00305474
Title: Identification and Treatment of the Liability to Develop Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: William Stone, PhD, Beth Israel- Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: XYMHI001
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
Keywords: Negative symptoms; neuropsychological deficits; Cognitive function; diagnostic; prevention
MeSH Terms: conditions — Schizophrenia; Disease | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Risperidone — Risperidone will be given in low dosage to a random sample of family members of Schizophrenic patients

SUMMARY:
This study seeks to determine whether adult, non-psychotic, first-degree relatives of schizophrenic patients who show specific neurocognitive deficits and negative symptoms will show improvements in these areas following a 6-month, double-blind trial of a low dose (up to 2.0 mg) of risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one first-degree biological relative with schizophrenia and their age is between 19 and 59.
* Desire to participate in a medication trial.
* Is able to provide informed consent.
* Having moderate levels of negative symptoms, defined as 6 items rated 3 or higher on the Scale for the Assessment of Negative Symptoms (SANS).
* Scoring two or more standard deviations below normal in at least one of three cognitive domains: vigilance/working memory, long-term verbal memory, and executive functions.
* Scoring at least one standard deviation below normal in a second cognitive domain.

Exclusion Criteria:

* IQ less than 80.
* Formal education less than 10 years.
* History of psychotic disorders.
* History of treatment with an antipsychotic medication.
* A substance abuse diagnosis within 6 months of diagnosis.
* A head injury with documented loss of consciousness exceeding 5 minutes (or subsequent cognitive deficits).
* A history of neurologic disease or damage.
* A medical condition with significant cognitive sequelae.
* A history of electroconvulsive treatment.

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-12; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological - cognitive measures | 2003-2010

SECONDARY OUTCOMES:
Psychiatric Symptoms | 2003-2010

CONTACTS AND LOCATIONS:
Overall Officials: William Stone, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Lingjiang Li, MD, PhD, Study Chair — Central South Unversity
Locations (1):
- Mental Health Institute, Changsha, Hunan, China